CLINICAL TRIAL: NCT00853073
Title: Does a New Add on (or Adjunctive) Therapy Used in Glaucoma Surgery Improve the Success of Needle Bleb Revisions?
Brief Title: Does Adding Bevacizumab Therapy in Glaucoma Surgery Improve the Success of Needle Bleb Revisions?
Acronym: Avastin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Marlene Moster, MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-867
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Glaucoma
Keywords: failing blebs; failing express shunt; avastin; bevacizumab; glaucoma; prior trabeculectomy; Express shunt placed under a scleral flap; subsequent filtration failure
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab; Hanks Balanced Salt Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab (Active Comparator): subjects will receive 1.0mg (0.04cc of 25 mg/ml) subconjunctival bevacizumab either temporal or nasal to the bleb following bleb needling procedure in addition to 0.1 cc mitomycin C.
  Interventions: Drug: bevacizumab
- balanced salt solution (Placebo Comparator): patients randomized to treatment B are given 0.04cc of balanced salt solution injected in identical fashion either temporal or nasal to the bleb following bleb needling procedure in addition to 0.1 cc mitomycin C.
  Interventions: Other: balanced salt solution

INTERVENTIONS:
Drug: bevacizumab — 1.0mg (0.04 cc of 25 mg/ml subconjunctival bevacizumab following bleb needling procedure
  Other Names: Avastin
  Arms: Bevacizumab
Other: balanced salt solution — 0.04 cc of balanced salt solution injected to the bleb following bleb needling procedure
  Arms: balanced salt solution

SUMMARY:
The purpose of this study is to see if a new add on (or adjunctive) therapy used in glaucoma surgery improves the success of needle bleb revisions.

DETAILED DESCRIPTION:
To investigate the efficacy of needle bleb revisions with mitomycin C with subconjunctival bevacizumab in promoting both filtering success and favorable bleb morphologic features.

ELIGIBILITY:
Inclusion Criteria:

* require glaucoma bleb needle revision with Mitomycin-C

Exclusion Criteria:

* pregnant, nursing, or not using adequate contraception
* other glaucoma eye surgery involving tube shunts
* prior retinal detachments surgery with scleral buckle
* infection, inflammation, or any abnormality preventing eye pressure measurement
* enrolled in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene R Moster, MD, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Institute, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tai TY, Moster MR, Pro MJ, Myers JS, Katz LJ. Needle bleb revision with bevacizumab and mitomycin C compared with mitomycin C alone for failing filtration blebs. J Glaucoma. 2015 Apr-May;24(4):311-5. doi: 10.1097/IJG.0b013e31829f9bd3. PMID 25826644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were recruited between February 2009 and July 2011 from the Glaucoma Service located at Wills Eye Hospital in Philadelphia.
Groups:
- Treatment A (Bevacizumab): patients randomized to treatment A are given 1.0mg (0.04cc of 25 mg/mL) subconjunctival bevacizumab injection either temporal or nasal to the bleb following bleb needling procedure in addition to 0.1 cc mitomycin C.
- Treatment B (Balanced Salt Solution): patients randomized to treatment B are given 0.04cc of balanced salt solution injected in identical fashion either temporal or nasal to the bleb following bleb needling procedure in addition to 0.1 cc mitomycin C.
Period: Overall Study
Arm/Group | Treatment A (Bevacizumab) | Treatment B (Balanced Salt Solution)
Started | 32 | 31
Completed | 29 | 29
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: 5 patients withdrew; 3 from Treatment A group and 2 from Treatment B group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A (Bevacizumab) | Treatment B (Balanced Salt Solution) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [37 to 91] | 71.2 [45 to 89] | 67.9 [37 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: mmHg (millimeters of mercury)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg (millimeters of mercury)
Arm/Group | Treatment A (Bevacizumab) | Treatment B (Balanced Salt Solution)
Number analyzed (Participants) | 29 | 29
mmHg (millimeters of mercury) | 11.52 [9.44 to 14.05] | 12.83 [10.44 to 15.77]

2. Secondary Outcome: Number of Participants With Surgical Success
Description: Surgery was rated as complete success, qualified success or failure. Complete success was defined as 20% (percent) reduction in eye pressure (IOP) without any IOP lowering medications. Qualified success was defined as 20% reduction of IOP with IOP lowering medications. Failure was defined as IOP greater than 21 mmHG (millimeters of mercury), less than 20% IOP reduction or need for additional surgery.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (Bevacizumab) | Treatment B (Balanced Salt Solution)
Number analyzed (Participants) | 29 | 29
Participants
  Complete success | 17 | 12
  Qualified success | 0 | 2
  Failure | 12 | 15

ADVERSE EVENTS:
Description: At each of the five post-operative follow-up visits, patients were assessed for visual acuity, intraocular pressure, anterior chamber depth, hypotony changes, endothelial folds, hyphema, flare, cells, optic nerve swelling, choroidal folds, choroidal detachment and macular/retina folds.
Arm/Group | Treatment A (Bevacizumab) | Treatment B (Balanced Salt Solution)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 17/29 | 15/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Bevacizumab) (N=29) | Treatment B (Balanced Salt Solution) (N=29)
Hyphema (Eye disorders) | 4 (4) | 3 (3)
Shallow Anterior Chamber (Eye disorders) | 7 (7) | 5 (5)
Shallow Anterior Chamber necessitating injection of viscoelastic (Eye disorders) | 1 (1) | 1 (1)
Endothelial folds (Eye disorders) | 4 (4) | 4 (4)
Retinal/Choroidal folds (Eye disorders) | 5 (5) | 5 (5)
Choroidals (Eye disorders) | 6 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size which did not allow further subgroup analysis based on these patient characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No